CLINICAL TRIAL: NCT00543673
Title: Tolerance of Healthy, Term Infants to Infant Formulas
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Abbott Nutrition (Industry)
Responsible Party: Bobbie Swearengin, Director Clinical Research Operations, Abbott Nutrition
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AK53
Record Dates: First submitted 2007-10-05; First posted 2007-10-15 (Estimated); Last update posted 2008-07-04 (Estimated); Status verified 2008-06

CONDITIONS: Healthy
Keywords: Healthy term infants
MeSH Terms: interventions — Milk, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Milk based formula A (Experimental): Experimental milk based infant formula
  Interventions: Other: Milk based formula A
- Standard formula (Active Comparator): standard milk based infant formula
  Interventions: Other: #2 Standard formula
- Reference (Other): Human milk
  Interventions: Other: #3 Human Milk
- Milk based formula C (Experimental): Experimental milk based infant formula
  Interventions: Other: Milk based formula C

INTERVENTIONS:
Other: Milk based formula A — feed as per HCP directions
  Other Names: AN0710A
  Arms: Milk based formula A
Other: #2 Standard formula — Feed as per HCP directions
  Other Names: AN0710B
  Arms: Standard formula
Other: #3 Human Milk — Feed as per HCP directions
  Other Names: Human Milk
  Arms: Reference
Other: Milk based formula C — Feed as per HCP direction
  Other Names: AN0710C
  Arms: Milk based formula C

SUMMARY:
To assess the gastrointestinal tolerance of healthy full-term infants fed either experimental formula or a control formula

ELIGIBILITY:
Inclusion Criteria:

* judged to be in good health.
* singleton from a full term birth with a gestational age of 37-42 weeks
* birth weight was > 2490 g (~5 lbs 8 oz)
* between 0 and 8 days of age at enrollment.
* Infant's parent(s) or a LAR has voluntarily signed and dated an ICF, approved by an Independent Ethics Committee/Institutional Review Board (IEC/IRB) and provided Health Insurance Portability and Accountability Act (HIPAA) (or other applicable privacy regulation) authorization prior to any participation in the study.

Exclusion Criteria:

* An adverse maternal, fetal or infant medical history thought by the investigator to have potential for effects on tolerance, growth, and/or development, including, but not limited to suspected maternal substance abuse.
* Infant has been treated with antibiotics.

Max Age: 8 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 180 (Actual)
Dates: Start 2007-09; Primary Completion 2008-05 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Mean rank stool consistency (MRSC) | Study Day 1 to Visit 3

SECONDARY OUTCOMES:
MRSC, percent watery stools, average number of stools per day, percent of feedings with spit-up and/or vomiting | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Timberly A. Williams, M.S., Study Chair — Abbott Nutrition, Abbott Laboratories
Locations (10):
- United States (10):
  - The Pediatric Clinic, North Little Rock, Arkansas
  - USF, Tampa, Florida
  - North Georgia Clinical Research, White's Pediatrics, Dalton, Georgia
  - Medical Associates Clinic, Dubuque, Iowa
  - Midwest Children's Health Research Institute, LLC, Lincoln, Nebraska
  - The Childrens Medical Group LLC, Poughkeepsie, New York
  - Levine Childrens Hospital, Charlotte, North Carolina
  - Ohio Pediatrics, Inc., Huber Heights, Ohio
  - Institute of Clinical Research, Mayfield Heights, Ohio
  - Scott & White Memorial Hospital, Temple, Texas

REFERENCES:
- [Derived] Williams T, Choe Y, Price P, Katz G, Suarez F, Paule C, Mackey A. Tolerance of formulas containing prebiotics in healthy, term infants. J Pediatr Gastroenterol Nutr. 2014 Nov;59(5):653-8. doi: 10.1097/MPG.0000000000000513. PMID 25061716